CLINICAL TRIAL: NCT03934320
Title: Improving Identification of Familial Hypercholesterolaemia in Primary Care Using a New Case Ascertainment Tool (FAMCAT)
Brief Title: Improving Identification of Familial Hypercholesterolaemia in Primary Care (FAMCAT)
Acronym: FAMCAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Nottingham (Other)
Collaborators: Newcastle University (Other); University College, London (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16090; 332 (Other Grant/Funding Number: NIHR School for Primary Care Research)
Record Dates: First submitted 2019-03-08; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAMCAT (Other)
  Interventions: Other: FAMCAT

INTERVENTIONS:
Other: FAMCAT — The intervention is a computer-based software algorithm (FAMCAT) for use in general practice with a family history questionnaire.

SUMMARY:
Multi-centre, non-randomised, non-controlled quasi-experimental study with nested qualitative study and economic appraisal.

Improving the identification of patients at high risk of cardiovascular disease in primary care, caused by conditions such as familial hypercholesterolaemia (FH), is a well-recognised national priority to prevent morbidity and mortality by early effective intervention.

This study will prospectively evaluate the clinical utility of the new primary care FH identification tool (FAMCAT) for identifying undiagnosed FH in routine primary care practice; and to assess its appropriateness, acceptability and cost-effectiveness.

This study will answer the following research questions (RQ):

1. What is the detection rate for new genetically-confirmed FH cases using the FAMCAT algorithm?
2. Is the FAMCAT tool appropriate and acceptable to practitioners and patients?
3. How can the FAMCAT tool be optimised to improve identification of FH?
4. What is the potential cost-effectiveness of the FAMCAT tool compared with current practice to identify patients with FH?
5. Can the FAMCAT intervention be improved?
6. What definitive study design and outcome measures are needed to provide robust evidence on whether to introduce FAMCAT into primary care practice?

RQ(1) & (3) will be answered by a quasi-experimental diagnostic accuracy study; RQ(2) & (5) answered by qualitative study; RQ (4) answered by economic appraisal and RQ(6) informed by all previous studies.

ELIGIBILITY:
Inclusion Criteria:

Patients - General practices

* Able to give written informed consent
* 18 years of age or over
* Serum cholesterol recorded in General Practice (GP) electronic records
* Registered with a participating GP practice
* Able to complete the self-administered questionnaires in English
* No previous recorded diagnosis of familial hypercholesterolaemia in their GP electronic health records
* Considered by their General Practitioner(s) to be appropriate to recruit to the study.

Patients - Secondary care

* Able to give written informed consent
* 18 years of age or over
* Referred to or under the care of participating Trusts (e.g. lipid clinics)
* Able to understand the study information and consent in English
* Considered by their healthcare professions to be appropriate to recruit to the study.

Staff

* Able to give written informed consent
* 18 years of age or over
* Working at a participating General Practice, Clinical Commissioning Group (CCG) or Secondary Care Trust.

Nominal Group

* Able to give written informed consent
* 18 years of age or over
* A FH stakeholder (including specialists, primary care commissioners, FH patient representative)

Exclusion Criteria:

Patients - General practices

* Unable to give written informed consent
* Under 18 years of age
* Serum cholesterol not recorded in GP electronic records
* Not registered with a participating GP practice
* Unable to complete the self-administered questionnaires in English
* Has a diagnosis of familial hypercholesterolaemia in their GP electronic records
* Unable to have a blood test (for medical or personal reasons)
* Have an opt-out code where patients has declined electronic medical records examined
* Considered by their General Practitioner(s) to be inappropriate to recruit due to psycho-social reasons, participating in another related clinical trial or significant health reasons, e.g. terminal illness/diagnosis.

Patients - Secondary care

* Unable to give written informed consent
* Under 18 years of age
* Not referred to or under the care of participating Trusts (e.g. lipid clinics)
* Unable to understand the study information and consent in English
* Considered by their healthcare professionals to be inappropriate to recruit to the study.

Staff

* Unable to give written informed consent
* Under 18 years of age
* Has not worked at a participating General Practice, CCG or Secondary Care Trust.

Nominal Group

* Unable to give written informed consent
* Under 18 years of age
* Not an FH stakeholder or FH patient representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Detection of genetically confirmed new FH cases using case identification tool (FAMCAT) | Through study completion, an average of 2 years
  Efficacy measure: Proportion (%) of genetically-confirmed FH cases Proportion (%) of genetically-confirmed FH cases

SECONDARY OUTCOMES:
Acceptability of FAMCAT | Through study completion, an average of 2 years.
  Efficacy measure: representativeness of qualitative interview sample. Key themes will be identified from qualitative interview transcripts of patient experience of participating in the study, acceptability of the study procedures (ie. location of blood test clinic appointments, waiting time to receive test results) , and appropriateness of methods of contact with study participants (ie. format and content of study materials, communicating test results). Key themes on usability will be identified from qualitative interview transcripts of health care professionals who used the FAMCAT tool clinically (ie. search criteria for clinical records, interpretation of results)
Appropriateness of FAMCAT | Through study completion, an average of 2 years.
  Efficacy measure: representativeness of qualitative interview sample. Key themes will be identified from qualitative interview transcripts of patient experience of appropriateness of methods of contact with study participants (ie. format and content of study materials, communicating test results).
Usability of FAMCAT | Through study completion, an average of 2 years.
  Efficacy measure: representativeness of qualitative interview sample. Key themes on usability will be identified from qualitative interview transcripts of health care professionals who used the FAMCAT tool clinically (ie. search criteria for clinical records, interpretation of results)
Self-reported anxiety measures for use in a future trial | Baseline to 15 months after genetic test results reported
  Anxiety measured using 6 item Spielberger State-Trait Anxiety Inventory (STAI). The total score will be calculated at study entry, after receiving genetic test results and 12- 15 months after genetic tests results received
Self-reported lifestyle change measures for use in a future trial | Baseline to 15 months after genetic test results reported
  Stages of change for smoking cessation and physical activity will be measured. The five stages of change will be dichotomised into: (1) pre-contemplation, contemplation and preparation and (2) action/maintenance. The distribution of proportions for each measure will be presented at study entry, after receiving genetic test results and 12- 15 months after genetic tests results received
Beliefs about predisposition to coronary heart disease | Baseline to 15 months after genetic test results reported
  Beliefs on causes for heart disease were assessed using 8 items, from a total of 18 items, which comprise the 'Causes of my illness' subscale in the Revised Illness Perception Questionnaire, IPQ-R.
  The distribution of data for each one of the 8 questions will be presented at study entry, after receiving genetic test results and 12- 15 months after genetic tests results received
Cost-effective FAMCAT threshold to identify genetically confirmed FH | through study completion, an average of 2 years
  Efficacy measure: Primary analysis:
  Incremental cost-effectiveness ratio (ICER) of FAMCAT compared to Simon-Broome criteria; Sensitivity analysis: Incremental costeffectiveness ratio (ICER) of FAMCAT at different testing thresholds. Short-term model: 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Qureshi, DM, Principal Investigator — University of Nottingham
Locations (1):
- Division of Primary Care, University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not have consent from participants to share their data for the purposes of future research.

REFERENCES:
- [Derived] Qureshi N, Akyea RK, Dutton B, Leonardi-Bee J, Humphries SE, Weng S, Kai J. Comparing the performance of the novel FAMCAT algorithms and established case-finding criteria for familial hypercholesterolaemia in primary care. Open Heart. 2021 Oct;8(2):e001752. doi: 10.1136/openhrt-2021-001752. PMID 34635577
- [Derived] Qureshi N, Akyea RK, Dutton B, Humphries SE, Abdul Hamid H, Condon L, Weng SF, Kai J; FAMCAT study. Case-finding and genetic testing for familial hypercholesterolaemia in primary care. Heart. 2021 Dec;107(24):1956-1961. doi: 10.1136/heartjnl-2021-319742. Epub 2021 Sep 14. PMID 34521694
- See also: Funder website — https://www.spcr.nihr.ac.uk/projects/improving-identification-of-familial-hypercholesterolaemia-in-primary-care-using-a-new-case-ascertainment-tool-famcat